CLINICAL TRIAL: NCT06808100
Title: Can Gdf-15 Level Predict Progression to Multiple Organ Failure in Patients With Septic Shock
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cihangir Doğu, Associate professor, Ankara City Hospital Bilkent
Other Study IDs: TABED 2-24-659
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Septic Shock; Multi Organ Failure
Keywords: Growth and differentiation factor 15; sepsis; septic shock; Multiple Organ Dysfunction Syndrome; Sequential Organ Failure Assessment score
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Blood sample for GDF-15 level at the day of admission
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group I: Patients older than 18 years of age who agreed to participate in the study. Patients fulfilling the inclusion criteria.
  Patients diagnosed with sepsis and in need of vasopressors. Patients treated in the intensive care unit for more than 48 hours.
  Patients whose blood sample could be collected for GDF-15 after transfer to the intensive care unit.

SUMMARY:
The aim of this observational study is to investigate whether GDF-15 levels can predict clinical outcome in patients admitted to the intensive care unit with a diagnosis of septic shock.

The main question is:

* Can the level of GDF-15 levels during ICU admission predict the development of multiple organ failure in patients with septic shock? All patients will continue to receive routine treatment for sepsis and septic shock. The investigators will observe the development of multiple organ failure by the Sequential Organ Failure Assessment (SOFA) score increase

DETAILED DESCRIPTION:
Sepsis can be defined as a disproportionate host response to infection. It has been reported that 2.8 million deaths per year in high-income countries are associated with sepsis. Excessive inflammatory response may lead to organ failure and death after multiple organ failure. After infection, pathogen-mediated molecular fragments (PAMPS) are formed and recognised by toll-like receptors and the immune system is activated. Pro- and anti-inflammatory mediators are released and levels of various cytokines increase. These changes affect neutrophil-endothelial adhesion, disrupt the coagulation cascade and increase microthrombi formation. The systemic inflammatory state may be followed by immune paralysis and secondary infections, which may lead to the loss of patients as a result of multiple organ failure.

Growth differentiation factor-15 (GDF-15), also known as macrophage inhibitory cytokine-1 (MIC-1), is a member of the transforming growth factor-β (TGFβ) superfamily. It is found in many tissues and is strongly expressed in epithelial cells and macrophages. Its level is correlated with macrophage activation. In recent years, circulating GDF-15 level has been identified as a biomarker with prognostic value in cardiopulmonary diseases such as heart failure myocardial infarction and pulmonary embolism. In addition, elevated GDF-15 levels have been shown in end-stage renal failure and acute respiratory distress syndrome and chronic inflammatory diseases.

Septic shock requires vasopressor support to maintain a mean arterial pressure of 65 mmHg despite adequate fluid replacement. Septic shock has a higher mortality rate and development of multiple organ failure is more common.

Although the correlation of elevated GDF-15 levels with organ failure has been shown, the relationship between GDF-15 levels and multiple organ failure in patients with septic shock has not yet been studied.

Primary aim in this study is to investigate the relationship between GDF-15 level measured after admission and progression to multiple organ failure in patients admitted to intensive care with septic shock.

Secondary aim is to predict mortality with GDF-15 level in patients treated in intensive care unit with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients older thab 18 years of age
* Patients with septic shock
* Patients without end-stage renal failure (KDIGO G4,G5)
* Patients without chronic liver disease
* Patients with New York Heart Association (NYHA) stage 1-2
* Patients not diagnosed with active cancer
* Non-pregnant patients
* Patients without chronic immunodeficiency
* Patients without chronic inflammatory disease

Exclusion Criteria:

* Patients younger than 18 years age
* Patients not diagnosed with septic shock
* Patients with end-stage renal failure
* Patients with chronic liver disease
* Patients with New York Heart Association (NYHA) stage 3-4
* Patients diagnosed with active cancer
* Pregnant patients
* Patients with chronic immunodeficiency
* Patients with chronic inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit of Ankara Bilkent City Hospital with a diagnosis of septic shock who met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Predicting the progression to multiple organ failure in patients admitted to intensive care unit with septic shock by GDF-15 level | Time from intensive care unit admission to mortality at the 28th day.
  Sequential Organ Failure Assessment (SOFA) score is a computational score used to assess the status of organ systems. The SOFA is based on six different scores scored from 0 to 4 for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems, with an increasing score reflecting worsening organ dysfunction. In the research, sepsis treatment and appropriate haemodynamic support treatment will be provided to patients and daily sofa score follow-up will be performed. Progression to multiple organ failure will be monitored with the sofa score.

SECONDARY OUTCOMES:
28-day intensive care mortality | 28 days after intensive care unit admission
  The GDF-15 level will be used to predict intensive care unit mortality within 28 days of intensive care unit admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In accordance with local legislation, the sharing of patient information is subject to special authorisation.